CLINICAL TRIAL: NCT03919955
Title: A Novel Pharmacological Therapy for Obstructive Sleep Apnea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Scott Aaron Sands, Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019P000666; R01HL146697 (NIH)
Record Dates: First submitted 2019-04-16; First posted 2019-04-18 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Atomoxetine Hydrochloride; oxybutynin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sequence A: Atomoxetine and Oxybutynin, then Placebo (Experimental): Sequence A: Atomoxetine and Oxybutynin, then Placebo
  Interventions: Drug: Atomoxetine; Drug: Oxybutynin; Drug: Placebo
- Sequence B: Placebo, then Atomoxetine and Oxybutynin (Experimental): Sequence B: Placebo, then Atomoxetine and Oxybutynin.
  Interventions: Drug: Atomoxetine; Drug: Oxybutynin; Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine — Atomoxetine 80 mg, per mouth, before bed. Participants will take the intervention nightly for one month. Half doses will be given on the first three nights.
  Other Names: Strattera
Drug: Oxybutynin — Oxybutynin 5 mg, per mouth, before bed. Participants will take the intervention nightly for one month. Half doses will be given on the first three nights.
  Other Names: Ditropan
Drug: Placebo — Placebo, per mouth, before bed.Participants will take the intervention nightly for one month. Half doses will be given on the first three nights.

SUMMARY:
A pharmacological, non-mechanical therapy for OSA that is efficacious and tolerable remains elusive. Here the investigators study the effect on sleep apnea severity of a combination of pharmacological agents (atomoxetine and oxybutynin, "AtoOxy") over a 1 month period of time. The current study will answer the following questions: Does ongoing, repeated-dose administration of atomoxetine-plus-oxybutynin (referred to as "AtoOxy") improve OSA severity, and do patients exhibit signs of symptomatic relief? Most importantly, which phenotypic subgroup of patients preferentially benefit from this intervention?

DETAILED DESCRIPTION:
Aim 1 - Effect of AtoOxy on sleep apnea severity. In a randomized controlled double-blind crossover study, 48 patients with moderate-to-severe OSA will take atomoxetine-plus-oxybutynin ("AtoOxy") versus placebo nightly for 1 month, with a 2-week washout in between. The investigators will test the hypothesis that AtoOxy reduces the Apnea-hypopnea index (primary outcome measure), and improves the following secondary outcomes:

* Nocturnal oxygenation, per "hypoxic burden of sleep apnea"
* Frequency of arousals from sleep (Arousal index)
* Self-reported sleepiness (Epworth Sleepiness Scale)
* Disease-specific quality of life (Functional Outcomes of Sleep Questionnaire, Short Form).
* Disease-specific quality of life (Sleep Apnea Quality of Life Index, Short Form)

Additional pre-specified exploratory outcome measures will be assessed, including Visual Analog Scales (Sleep Quality, Treatment Satisfaction) and additional polysomnographic measures of sleep (Stage 1 sleep, %total sleep time). Adherence and adverse events will also be carefully monitored to assess repeated-dose tolerance of the intervention.

Aim 2 - Determine which patient phenotypes respond best to AtoOxy. Patients will also take part in an additional night before initiating study medication to measure the key mechanisms causing OSA. The investigators will prospectively test the hypothesis that greater pharyngeal collapsibility determines a reduced response to therapy. They will also separately test the hypotheses that a reduced muscle responsiveness, reduced baseline muscle activation, a higher arousal threshold, and a lower loop gain will facilitate a greater response to therapy.

ELIGIBILITY:
Inclusion criteria:

* Ages 21-70 years
* Diagnosed OSA or clinically-suspected OSA
* Not using CPAP (>1 month).

Exclusion criteria:

* Any uncontrolled medical condition
* Current use of the medications under investigation
* Use of medications expected to stimulate or depress respiration (including opioids, barbiturates, doxapram, almitrine, theophylline, 4-hydroxybutanoic acid).
* Current use of hypnotic medications (trazodone, eszopiclone, benzodiazepines).
* Current use of SNRIs/SSRIs or anticholinergic medications.
* Conditions likely to affect obstructive sleep apnea physiology: neuromuscular disease or other major neurological disorder, heart failure (also below), or any other unstable major medical condition.
* Respiratory disorders other than sleep disordered breathing:

chronic hypoventilation/hypoxemia (awake SaO2 < 92% by oximetry) due to chronic obstructive pulmonary disease or other respiratory conditions.

* Other sleep disorders: periodic limb movements (periodic limb movement arousal index > 10/hr), narcolepsy, or parasomnias.
* Contraindications for atomoxetine and oxybutynin, including:

  * hypersensitivity to study drugs (angioedema or urticaria)
  * pheochromocytoma
  * use of monoamine oxidase inhibitors
  * benign prostatic hypertrophy, urinary retention
  * untreated narrow angle glaucoma
  * bipolar disorder, mania, psychosis
  * history of major depressive disorder (age<24).
  * history of attempted suicide or suicidal ideation within one year prior to screening
  * clinically significant constipation, gastric retention
  * pre-existing seizure disorders
  * clinically-significant kidney disorders (eGFR<60 ml/min/1.73m2)
  * clinically-significant liver disorders
  * clinically-significant cardiovascular conditions
  * severe hypertension (SBP>180 mmHg or DBP>110 mmHg measured at baseline)
  * cardiomyopathy (LVEF<50%) or heart failure
  * advanced atherosclerosis
  * history of cerebrovascular events
  * history of cardiac arrhythmias e.g., atrial fibrillation, QT prolongation
  * other serious cardiac conditions that would raise the consequences of an increase in blood pressure or heart rate
  * myasthenia gravis
  * pregnancy/breast-feeding
* Allergy to lidocaine (Aim 2 only)
* Claustrophobia
* Pregnancy or nursing

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Sands, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected during the study, after deidentification, will be available 12 months after publication to researchers who provide a methodologically sound proposal for any purpose.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately after publication. No end date.
Access Criteria: 1-page proposals should be directed to Dr. Scott Sands (sasands@bwh.harvard.edu). To gain access, requestors will be asked to sign a data use agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 117 were enrolled, 58 passed baseline screening and were randomized.
Groups:
- Sequence AB; Sequence BA: Patients randomized to Placebo then Active
Period: Overall Study
Arm/Group | Sequence AB | Sequence BA
Started | 29 | 29
Completed Treatment Period 1 | 26 | 27
Started Treatment Period 2 | 26 | 26
Completed | 26 | 24
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- All Participants: All participants
Arm/Group | All Participants
Number analyzed (Participants) | 58
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 52 [41 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 35
  More than one race | 2
  Unknown or Not Reported | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 50
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Apnea-hypopnea Index [AHI]
Description: Apneas and hypopneas per hour (3% desat and/or arousal), % change from baseline
Time Frame: one month
Population: Population reported here is the population who completed a given treatment period. (Rather, formal statistical analysis was performed using multiple imputation.)
Measure: Median (Inter-Quartile Range); unit: events/hr; % change from baseline
Groups:
- Active Intervention: Active Intervention
- Placebo Intervention: Placebo intervention
Arm/Group | Active Intervention | Placebo Intervention
Number analyzed (Participants) | 50 | 53
events/hr; % change from baseline | -11.8 [-44.9 to 7.2] | -2.3 [-29.3 to 17.6]

2. Secondary Outcome: Hypoxic Burden
Description: Desaturation area under curve × event frequency, % change from baseline
Time Frame: one month
Population: secondary outcomes are presented as per primary outcome
Measure: Median (Inter-Quartile Range); unit: %.min/hr; % change from baseline
Arm/Group | Active Intervention | Placebo Intervention
Number analyzed (Participants) | 50 | 53
%.min/hr; % change from baseline | -15.0 [-46.9 to 22.3] | -8.7 [-26.9 to 19.9]

3. Secondary Outcome: Arousal Index
Description: Scored EEG arousals per hour (>3 s), % change from baseline
Time Frame: one month
Measure: Median (Inter-Quartile Range); unit: events/hr; % change from baseline
Arm/Group | Active Intervention | Placebo Intervention
Number analyzed (Participants) | 50 | 53
events/hr; % change from baseline | -0.3 [-23.9 to 41.5] | -3.7 [-26.2 to 22.2]

4. Secondary Outcome: Epworth Sleepiness Scale
Description: Self-reported sleepiness on scale of 0-24, higher values indicated greater sleepiness
Time Frame: one month
Population: All participants who completed questionnaires on treatment.
Measure: Median (Inter-Quartile Range); unit: units on a scale; change from baseline
Arm/Group | Active Intervention | Placebo Intervention
Number analyzed (Participants) | 51 | 53
units on a scale; change from baseline | 0 [-3 to 2] | -1 [-3 to 2]

5. Secondary Outcome: Functional Outcomes of Sleep Questionnaire, Short Form
Description: Disease-specific daytime function on scale of 5-20, higher values indicate greater function and quality of life
Time Frame: one month
Measure: Median (Inter-Quartile Range); unit: units on a scale; change from baseline
Arm/Group | Active Intervention | Placebo Intervention
Number analyzed (Participants) | 51 | 53
units on a scale; change from baseline | 0.33 [-1.0 to 1.5] | 0 [-1.0 to 2.0]

6. Secondary Outcome: Sleep Apnea Quality of Life Index, Short Form
Description: Disease-specific quality of life on scale of 1-7, higher values indicate greater sleep-apnea related quality of life
Time Frame: one month
Measure: Median (Inter-Quartile Range); unit: units on a scale; change from baseline
Arm/Group | Active Intervention | Placebo Intervention
Number analyzed (Participants) | 51 | 53
units on a scale; change from baseline | 0.3 [-0.1 to 1.0] | 0.4 [0 to 1.1]

ADVERSE EVENTS:
Time Frame: One month
Description: Systematically documented per checklist, plus additional space to note new AEs. Subclassified as mild, moderate, or severe by self-report.
Arm/Group | Active Intervention | Placebo Intervention
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 1/55 | 0/55
Other Adverse Events (participants affected / at risk) | 39/55 | 20/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Intervention (N=55) | Placebo Intervention (N=55)
Hospitalization and laparotomy for suspected bowel obstruction (Gastrointestinal disorders) | 1 | 0 — Bowel obstruction not confirmed by laparotomy procedure; SAE reviewed by the DSMB and determined to be <50% likelihood of being related to the study intervention.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Intervention (N=55) | Placebo Intervention (N=55)
Dry mouth (Gastrointestinal disorders) | 27 | 11 — moderate-to-severe
Drowsiness/Fatigue (General disorders) | 13 | 8 — moderate-to-severe
Insomnia (General disorders) | 13 | 2 — moderate-to-severe
Decreased appetite (Gastrointestinal disorders) | 8 | 1
Restlessness (General disorders) | 8 | 1 — moderate-to-severe
Constipation (Gastrointestinal disorders) | 8 | 0 — moderate-to-severe
Nausea (Gastrointestinal disorders) | 7 | 2 — moderate-to-severe
Dificulty urinating (General disorders) | 6 | 1 — moderate-to-severe
Sexual problems / decreased libido (General disorders) | 6 | 0 — moderate-to-severe
Abdominal discomfort / pain (Gastrointestinal disorders) | 5 | 1 — moderate-to-severe
Dry skin (General disorders) | 4 | 1 — moderate-to-severe
Headache (General disorders) | 4 | 1 — moderate-to-severe
Indigestion (Gastrointestinal disorders) | 4 | 0 — moderate-to-severe
Dizziness (Ear and labyrinth disorders) | 3 | 1 — moderate-to-severe
Erectile dysfunction (General disorders) | 3 | 0 — moderate-to-severe
Vomiting (Gastrointestinal disorders) | 3 | 0 — moderate-to-severe
Difficulty swallowing (Gastrointestinal disorders) | 3 | 0 — moderate-to-severe

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT03919955/Prot_SAP_000.pdf